CLINICAL TRIAL: NCT01173289
Title: A Phase II Study of External Beam Radiotherapy for Locoregionally Advanced or Recurrent Differentiated Thyroid Carcinoma
Brief Title: Study of External Beam Radiotherapy to Thyroid Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Tae Hyun Kim, Principal Investigator, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-09-436
Record Dates: First submitted 2010-07-22; First posted 2010-08-02 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Thyroid Cancer
Keywords: Thyroid Carcinoma; External Beam Radiotherapy
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- External Beam Radiotherapy (Experimental): Definition of target volume:
  * Gross tumor volume (GTV) = gross tumor defined with intravenous bolus contrast administration given CT scan
  * Clinical target volume (CTV) = GTV + included volumes of clinical and suspected subclinical involvement (draining lymph nodes)
  * Planning target volume (PTV) = CTV + 5-10 mm of lateral, craniocaudal, and anteroposterior margins.
  Radiation dose and planning :
  * Total dose 65 Gy for gross tumor, 62.4 Gy for microscopic involved area, 58.5 Gy for high risk lymph node area and 52 Gy for elective lymph node area in 26 fractions during 6 weeks
  * Dose prescription: 90% isodose volume of prescribed dose encompassed PTV
  * The dose-volume histogram (DVH) of targets, such as GTV, CTV, and PTV, and the normal tissues, such as the esophagus, lung, contralateral normal thyroid, arytenoids, vocal cord and spinal cord, etc., was calculated.
  Interventions: Radiation: External Beam Radiotherapy

INTERVENTIONS:
Radiation: External Beam Radiotherapy — Definition of target volume:
  * Gross tumor volume (GTV) = gross tumor defined with intravenous bolus contrast administration given CT scan
  * Clinical target volume (CTV) = GTV + included volumes of clinical and suspected subclinical involvement (draining lymph nodes)
  * Planning target volume (PTV) = CTV + 5-10 mm of lateral, craniocaudal, and anteroposterior margins.
  Radiation dose and planning
  * Total dose 65 Gy for gross tumor, 62.4 Gy for microscopic involved area, 58.5 Gy for high risk lymph node area and 52 Gy for elective lymph node area in 26 fractions during 6 weeks
  * Dose prescription: 90% isodose volume of prescribed dose encompassed PTV
  * The dose-volume histogram (DVH) of targets, such as GTV, CTV, and PTV, and the normal tissues, such as the esophagus, lung, contralateral normal thyroid, arytenoids, vocal cord and spinal cord, etc., was calculated.

SUMMARY:
The primary objective of this study is to estimate the 5 year locoregional control rate after External Beam Radiotherapy (EBRT) in the patient with locally advanced differentiated thyroid cancer. In a prior retrospective trial for this same group of patients, the 5 year locoregional control rate was 85% in EBRT group and 70% in no EBRT group. For the total number of patients to detect a minimum of 20% improvement in 5 year locoregional control rate with 80% of statistical power and the 5% significance level, the table for sample size planning given by Makuch and Simon was chosen. Forty-three patients are required for this regimen to regard as worthy of further investigation. Considering 15% follow up loss, 50 eligible patients will be enrolled.

DETAILED DESCRIPTION:
The standard approaches to the treatment of differentiated thyroid cancer include surgical resection, radioactive iodine treatment, and thyroid-stimulating hormone suppression. The role of external beam radiotherapy (EBRT), however, remains controversial.

The purpose of this phase II study is to evaluate the impact of EBRT on the locoregional control in locoregionally advanced or recurrent differentiated thyroid cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed differentiated thyroid cancer
* Patient with locally advanced tumor (T4a, tumor of any size extending beyond the thyroid capsule to invade subcutaneous soft tissues, larynx, trachea, esophagus, or recurrent laryngeal nerve or T4b, tumor invades prevertebral fascia or encases carotid artery or mediastinal vessels or N1b, unilateral, bilateral, or contralateral cervical or mediastinal lymph node positive), or locoregionally recurrent tumor
* All patients must have radiographically assessable disease
* No previous irradiation to the planned field
* Age of ≥ 18 years
* Performance status of 0 to 2 on the Eastern Cooperative Oncology Group (ECOG) score
* Required Entry Laboratory Parameters WBC count ≥ 1,000/mm3; hemoglobin level ≥ 7.5 g/dL; platelet count ≥ 100,000/mm3; creatinine ≤ 3.0 mg/dL
* Oral intake (including J-tube feeding) of ≥ 1,500 calories/day should be maintained.
* Signed informed consent form prior to study entry

Exclusion Criteria:

* Patient with anaplastic carcinoma (focal anaplastic change associate with differentiated thyroid cancer is not excluded)
* Age of <18 years
* Previous history of RT adjacent to planned field
* Poor performance status of 3 to 4 on the Eastern Cooperative Oncology Group (ECOG) score
* Pregnant or breast feeding status
* Previous history of uncontrolled other malignancies within 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2009-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
All cause mortality | Two Years

CONTACTS AND LOCATIONS:
Overall Officials: Tea Hyun Kim, M.D., Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Korea, Goyang-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Lee EK, Lee YJ, Jung YS, Ryu J, Kim TH, Lee CY, Ryu CH, Kim TS, Kim SK, Chung KW, Kim SS, Kim DY, Kim JY, Cho KH. Postoperative simultaneous integrated boost-intensity modulated radiation therapy for patients with locoregionally advanced papillary thyroid carcinoma: preliminary results of a phase II trial and propensity score analysis. J Clin Endocrinol Metab. 2015 Mar;100(3):1009-17. doi: 10.1210/jc.2014-3242. Epub 2015 Jan 12. PMID 25581596